CLINICAL TRIAL: NCT03169712
Title: Efficacy of Sequential Imagery Rehearsal Therapy and Cognitive-Behavioural Therapy in Sexual Assault Victims With Posttraumatic Stress Disorder: a Randomized Control Trial
Brief Title: IRT and CBT in Sexual Assault Victims With PTSD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Laval University (Other)
Responsible Party: Principal Investigator, Geneviève Belleville, Associate Professor, Laval University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 000000
Record Dates: First submitted 2017-05-23; First posted 2017-05-30 (Actual); Last update posted 2023-10-06 (Actual); Status verified 2023-10

CONDITIONS: Stress Disorders, Post-Traumatic
MeSH Terms: conditions — Stress Disorders, Post-Traumatic | interventions — Cognitive Behavioral Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- CBT for PTSD (Active Comparator): 15 sessions of trauma-focused CBT
  Interventions: Behavioral: Cognitive Behavioral Therapy for PTSD
- Imagery Rehearsal Therapy + CBT for PTSD (Experimental): 5 sessions of IRT + 15 sessions of trauma-focused CBT
  Interventions: Behavioral: Cognitive Behavioral Therapy for PTSD; Behavioral: Imagery Rehearsal Therapy

INTERVENTIONS:
Behavioral: Cognitive Behavioral Therapy for PTSD — Trauma-focused CBT protocol elaborated by Marchand and Guay from the Trauma Studies Centre at Louis-H. Lafontaine Hospital in Montreal and adapted from Foa, Hembree and Rothbaum (2007)
Behavioral: Imagery Rehearsal Therapy — IRT protocol published by Nappi and collaborators (2010)
  Arms: Imagery Rehearsal Therapy + CBT for PTSD

SUMMARY:
Sexual assault victims (SAV) have an elevated risk of developing posttraumatic stress disorder (PTSD). Trauma-focused cognitive-behavioural therapy (CBT) is an effective first-line treatment for this pathology. However, although sleep disturbances are a common complaint in SAV with PTSD, trauma-focused CBT does not directly address this symptom. Posttraumatic nightmares are widespread among SAV. Trauma-related sleep disturbances are associated with significant impairment in general functioning and quality of life (mental and physical health), and contribute to the maintenance of PTSD symptoms. This study evaluates the efficacy of sequential nightmare therapy (imagery rehearsal therapy; IRT) and trauma-focused CBT, in comparison to CBT alone. Forty-two SAV suffering from PTSD and sleep difficulties were recruited and randomly assigned to the experimental (IRT+CBT) or control condition (waiting period followed by CBT alone). Participants were administered a clinical interview and a series of questionnaires assessing PTSD symptoms, general functioning and quality of life.

ELIGIBILITY:
Inclusion Criteria:

* over 18 years of age;
* able to understand and speak French;
* history of unwanted sexual experience;
* PTSD diagnosis according to DSM-IV-TR;
* sleep complaints, as established by Pittsburgh Sleep Quality Index score ≥ 5 and a mean of one or more NM per week for at least one month;
* if psychotropic medication was used, (antidepressant, antianxiety, antipsychotic or hypnotic medication) stable for a minimum of three months;
* available for in-person assessments and therapy sessions.

Exclusion Criteria:

* past or present psychotic episode, bipolar disorder or organic mental disorder (e.g. dementia);
* substance use disorder;
* sleep apnea diagnosis;
* use of prazosine to treat nightmares;
* presently in treatment for psychological difficulties;
* significant suicidal thoughts requiring immediate intervention.

Ages: 18 Years to 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 42 (Actual)
Dates: Start 2012-12-20 (Actual); Primary Completion 2016-05-01 (Actual); Study Completion 2016-08-01 (Actual)

PRIMARY OUTCOMES:
Change in Pittsburgh Sleep Quality Index total score | Pre-Treatment; Post-Treatment 1 (5 weeks after pre-treatment); Post-Treatment 2 (20 weeks after pre-treatment); 3-month FU; 6-month FU; 12-month FU
  Self-report questionnaire
Change in Modified PTSD Symptom Scale - Self Report total score | Pre-Treatment; Post-Treatment 1 (5 weeks after pre-treatment); Post-Treatment 2 (20 weeks after pre-treatment); 3-month FU; 6-month FU; 12-month FU
  Self-report questionnaire

SECONDARY OUTCOMES:
Change in Nightmare Distress Questionnaire total score | Pre-Treatment; Post-Treatment 1 (5 weeks after pre-treatment); Post-Treatment 2 (20 weeks after pre-treatment); 3-month FU; 6-month FU; 12-month FU
  Self-report questionnaire
Change in Pittsburgh Sleep Quality Index - Addendum for PTSD total score | Pre-Treatment; Post-Treatment 1 (5 weeks after pre-treatment); Post-Treatment 2 (20 weeks after pre-treatment); 3-month FU; 6-month FU; 12-month FU
  Self-report questionnaire
Change in World Health Organization Disability Assessment Schedule total and subscale scores | Pre-Treatment; Post-Treatment 1 (5 weeks after pre-treatment); Post-Treatment 2 (20 weeks after pre-treatment); 3-month FU; 6-month FU; 12-month FU
  Self-report questionnaire
Change in Medical Outcomes Study Health Survey subscale scores | Pre-Treatment; Post-Treatment 1 (5 weeks after pre-treatment); Post-Treatment 2 (20 weeks after pre-treatment); 3-month FU; 6-month FU; 12-month FU
  Self-report questionnaire
Change in Beliefs About Psychological Service total score | Pre-Treatment; Post-Treatment 1 (5 weeks after pre-treatment); Post-Treatment 2 (20 weeks after pre-treatment); 3-month FU; 6-month FU; 12-month FU
  Self-report questionnaire
Change in Working Alliance Inventory subscale scores | Pre-Treatment; Post-Treatment 1 (5 weeks after pre-treatment); Post-Treatment 2 (20 weeks after pre-treatment); 3-month FU; 6-month FU; 12-month FU
  Self-report questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: Geneviève Belleville, Principal Investigator — Laval University
Locations (1):
- Service de Consultation de l'École de Psychologie, Québec, Quebec, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] O'Doherty L, Whelan M, Carter GJ, Brown K, Tarzia L, Hegarty K, Feder G, Brown SJ. Psychosocial interventions for survivors of rape and sexual assault experienced during adulthood. Cochrane Database Syst Rev. 2023 Oct 5;10(10):CD013456. doi: 10.1002/14651858.CD013456.pub2. PMID 37795783
- [Derived] Belleville G, Dube-Frenette M, Rousseau A. Efficacy of Imagery Rehearsal Therapy and Cognitive Behavioral Therapy in Sexual Assault Victims With Posttraumatic Stress Disorder: A Randomized Controlled Trial. J Trauma Stress. 2018 Aug;31(4):591-601. doi: 10.1002/jts.22306. Epub 2018 Aug 2. PMID 30070398